CLINICAL TRIAL: NCT00299390
Title: Phase II Study to Investigate the Efficacy and Safety of ZK 219477 as First Line Therapy in Chemotherapy Naive Patients With Extensive Disease (ED) Stage Small Cell Lung Cancer (SCLC)
Brief Title: Safety and Efficacy Study of a New Chemotherapy Agent to Treat Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Since only 1 of the first 10 subjects responded to the study treatment, it was decided to stop the trial due to lack of efficacy .
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 91375; 2005-000597-53 (EudraCT Number); 307972
Record Dates: First submitted 2006-03-03; First posted 2006-03-06 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Small Cell Lung Carcinoma
Keywords: Sagopilone; Epothilone; SCLC; Small Cell Lung Cancer; Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms | interventions — sagopilone

ARMS (1):
- Sagopilone (Experimental)
  Interventions: Drug: Sagopilone (BAY86-5302, ZK 219477)

INTERVENTIONS:
Drug: Sagopilone (BAY86-5302, ZK 219477) — Sagopilone; 16 mg/m2 (maximum 32 mg) as 3 hour i.v. infusion

SUMMARY:
The purpose of this study is to determine whether the study drug is effective and safe in the first line treatment of patients with small cell lung cancer

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven Small-cell lung cancer (SCLC)
* Stage of extensive disease defined by the presence of distant metastases
* At least 1 unidimensionally measureable lesion
* WHO performance status 0 to 1
* No previous SCLC-related chemotherapy
* No previous SCLC-related surgery
* No previous radiotherapy (excepting for brain metastasis)
* Adequate function of major organs and systems

  * Nervous system

    * No Grade 2 or greater peripheral neuropathy
  * Cardiovascular:

    * No symptomatic congestive heart failure
    * No unstable angina pectoris
    * No arrythmia needing continuous treatment
    * No other uncontrolled concurrent illness

Exclusion Criteria:

* Superior vena cava syndrome or obstruction of any vital structure
* Untreated malignant hypercalcemia
* Pleural effusion as the only manifestation of disease
* Extensive disease amenable to radiation therapy
* Symptomatic brain metastases requiring whole brain irradiation
* Any concomitant malignancy excepting non-melanoma skin cancer or carcinoma in situ of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-04; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Response to treatment according to the modRECIST (complete response or partial response) | Every 2 cycles until tumor progression i.e. approximately every 6 weeks

SECONDARY OUTCOMES:
Duration of complete or partial tumor response | Every 2 cycles until tumor progression i.e. approximately every 6 weeks
Time to tumor progression | Every 2 cycles until tumor progression i.e. approximately every 6 weeks
Number of participants with adverse events | Approximately 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/